CLINICAL TRIAL: NCT02359812
Title: Robot-Aided Diagnosis, Passive-Active Arm Motor and Sensory Rehabilitation Post Stroke: Aim 1
Brief Title: Robot Aided Rehabilitation - Multi-joint Evaluations
Acronym: Aim1
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); North Carolina State University (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00074975
Record Dates: First submitted 2015-01-23; First posted 2015-02-10 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Upper extremity; Rehabilitation; Robot; Hemiplegia; Spasticity; Arm; Hand
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy volunteers with no history of neurological disorders
- Stroke: Patients had a recent stroke, two weeks or earlier prior to enrollment

SUMMARY:
Sensory and motor impairments following stroke can lead to substantial disability involving the arm and hand. The investigator hypothesized that excessive local and cross-coupled stiffness, diminished individuation and proprioceptive acuity will be present among multiple degree of freedom in the upper limb. The stiffness and spasticity will increase with time post-stroke. The objective of this study is to quantify the progression throughout the arm and hand during recovery from stroke. The investigator will measure the clinical assessment scores, and neuromechanical properties including range of motion, active and passive cross coupling, and spasticity by the IntelliArm robot.

DETAILED DESCRIPTION:
Sensorimotor impairments following stroke can lead to substantial disability involving the upper extremity. These impairments often involve complex pathological changes across multiple joints and multiple degrees of freedom of the arm and hand, thereby rendering them difficult to diagnose and treat. Many potential mechanisms, such as muscle weakness, motoneuronal hyperexcitability, and elevated passive joint impedance, can contribute to the impairments, thereby making it difficult to discern where best to focus treatment.

Objectives: The objectives of this study are to quantify the progression of neuromechanical properties throughout the upper extremity during recovery from stroke.

Specific Aim 1: The specific aim is to examine neuromechanical properties throughout the entire upper extremity and corticomotor excitability in stroke survivors over a period of 6 months and throughout the progression from the acute to the subacute to the chronic phases of recovery.

Hypothesis: Excessive local and cross-coupled stiffness, heteronymous reflexes, corticomotor excitability, and diminished individuation and proprioceptive acuity will be present among multiple degree of freedom in the upper limb. The stiffness and spasticity will increase with time post-stroke.

The aim of this study will be addressed through a longitudinal evaluation of stroke survivors over the first 6 months following the stroke. Specifically, upper extremity control and neuromechanical properties will be measured at 7 different time points over the six months.

36 stroke survivors from 18-85 years old will be recruited over the duration of the study. A group of 20 healthy subjects will be recruited to obtain the normal values of the neuromuscular and biomechanical properties.

In an initial screening session, after the subject has consented, a research personnel will check the subject's health status and conduct clinical examinations in order to determine if the subject meets the inclusion and exclusion criteria. During the screening session, the subject will participate in several clinical assessments. The screening evaluations will take about one half hour.

If the subject qualifies for the study, the subject will participate in evaluation sessions at 7 time points spaced throughout the study. For each evaluation session, participants will be asked to come to our laboratories. Evaluation of participants will have neuromechanical and clinical components. The neuromechanical components of the evaluation will take approximately 3 hours, and the clinical evaluation will need about 2.5 hours.

Neuromechanical evaluations: In diagnosing the multi-joint and multi-degree of freedom (DOF) neuromechanical changes at the upper impaired limb, the IntelliArm will operate both passive and active modes. During neuromechanical evaluations, the subject will sit upright on a barber's chair and the trunk will be strapped to the backrest of the chair. The subject's arm, forearm and hand will be strapped to the corresponding braces which are attached on the robotic arm. The relevant servomotor-axles of the IntelliArm are aligned with the subject's arm at the shoulder, elbow, wrist, and metacarpophalangeal (MCP) joints. The adjustments will be made for the robotic arm to work properly with each subject.

Electromyography (EMG) system may be employed for recording the muscle activities at the upper impaired limb. The skin over the muscle belly will be cleaned with an alcohol pad and may be shaved by disposable razors. Self-adhesive electrodes will be placed on the cleaned sites and connected to the instrument and computer. The surface electrodes may be put on several different muscle bellies, including Flexor digitorum superficialis (FDS), Extensor digitorum (ED), Flexor carpi radialis (FCR), Extensor carpi radialis longus (ECRL), Biceps Brachii (BB), Triceps Brachii long head (TBLH), Deltoid anterior (DA), and Deltoid posterior (DP).

After all preparations are made, the evaluation will begin with the passive movement first. In the passive mode, the multi-joint arm robot will move the shoulder, elbow, wrist and fingers of the impaired arm of stroke survivors throughout the ROMs both simultaneously and individually in well-controlled spatial and temporal patterns with multi-axis torques and positions measured at the shoulder, elbow, wrist and MCP joints. Those joints will be moved one at a time or all of them will be moved together randomly, and the movements will be repeated for up to 5 times in each condition. After finishing the evaluation of passive motion, the participant will randomly be asked to move each joint of the upper limb or move the whole upper limb from one place to another, and will need each participant to repeating the movement for up to 5 times in each condition. Each neuromechanical evaluation will take approximately 3 hours.

The joint torque and angular displacement of each joint will be recorded. During the evaluation sessions, participant's reflex responses and muscle activities, such as hyperexcitability of the flexors and voluntary contractions of agonist and antagonist muscles at each joint, will be recorded and monitored through the skin electrodes with wireless EMG system. The electrodes are just used for recording the signal generated by the muscles and the participant will not feel any shocks during the evaluations. Non-invasive electroencephalography (EEG) electrodes may be attached on the scalp to record brain activity signals. A video or some photos may be taken as an option to evaluate the movement patterns during the evaluations.

Measures of stiffness and of hyperexcitability of the finger/wrist flexor muscles, namely spasticity and relaxation time, will also be made using techniques investigators have implemented successfully in the past. Spasticity of wrist/hand muscles will be measured as the reflex response to imposed rotation of the wrist joint. A servomotor will create either fast wrist rotation to invoke a stretch reflex or slow constant-velocity rotation to measure nominally passive stiffness. Wrist angle, angular velocity, and torque are recorded for analysis of spasticity. EMG recordings will be obtained with surface electrodes from selected superficial muscles. Relaxation time will be quantified by examining flexor muscle activity. The subject will be instructed to grip maximally upon hearing an audible tone. The subject should then relax the grip as quickly as possible after hearing a second tone. The relaxation time is defined as elapsed time from the second tone to the point at which the flexor muscle magnitude returns to the baseline level + three standard deviations.

Clinical evaluations: During clinical evaluations subjects will undergo a battery of standardized clinical assessments. These assessments require subjects to complete functional movements and tasks using the arms and hands. The clinical assessments to be administered include those listed below.

Screening Mini Mental State Exam Chedoke McMaster Stroke Assessment: Impairment Inventory of Arm and Hand

Full Evaluation Sessions Graded Wolf Motor Function Test (WMFT) Fugl-Meyer Upper Extremity (FMUE) Chedoke McMaster Stroke Assessment: Impairment Inventory of Arm and Hand Action Research Arm Test (ARAT) Nottingham Sensory Assessment Modified Ashworth Scale (MAS) Grip Strength & Pinch Strength

ELIGIBILITY:
Inclusion Criteria:

1. First focal unilateral lesion, ischemic or hemorrhagic
2. Had a stroke less than a month prior to enrollment
3. Rated between stages 1-4 on the Chedoke McMaster Stroke Assessment Impairment Inventory: Stage of Recovery of the Arm
4. Rated between stages 1-4 on the Chedoke McMaster Stroke Assessment Impairment Inventory: Stage of Recovery of the Hand

Exclusion Criteria:

1. Apraxia
2. Other unrelated or musculoskeletal injuries
3. Unable to sit in a chair for 3 consecutive hours
4. Score of less than 22 on the Mini Mental Status Exam
5. Poor fit into equipment used in study which compromises proper use. This will be determined by the judgment of study staff

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients at a rehabilitation hospital, patients at an acute care hospital, patients from outpatient clinics, patients from day rehabilitation programs.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Graded Wolf Motor Function Test (WMFT) at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The WMFT is a quantitative measure of upper extremity motor ability through timed and functional tasks.

SECONDARY OUTCOMES:
Changes from baseline Fugl-Meyer Upper Extremity at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Changes from baseline Chedoke McMaster Stroke Assessment: Impairment Inventory of Arm and Hand at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The Chedoke-McMaster Stroke Assessment (CMSA) is a screening and assessment tool utilized to measure physical impairment and activity of an individual following a stroke. The Chedoke Arm and Hand Activity Inventory (CAHAI) is used to assess functional ability of the paretic arm and hand. Each domain is scored on a 7-point scale.
Changes from baseline Modified Ashworth Scale (MAS) at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Changes from baseline Action Research Arm Test (ARAT) at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  ARAT assesses the ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Changes from baseline Grip Strength & Pinch Strength at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  A dynamometer is used to measure grip strength and a pinch gauge to measure tip, key, and palmar pinch.
Changes from baseline Nottingham Sensory Assessment at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The assessment tests the tactile sensation of the patient through light touch, pressure and pinprick.
Changes from baseline Range of motion (ROM) at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  The range of motion (ROM) of shoulder, elbow, wrist and fingers will be measured in Degree.
Changes from baseline spasticity at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  Spasticity will be measured by the resistance torque in Newton-meter under controlled movement at each joint.
Changes from baseline relaxation time of the finger flexor muscles at six time points | 2 week (baseline), 1 month, 2 month, 3 month, 4 month, 5 month and 6 month post stroke
  Relaxation time will be quantified in Second by examining flexor muscle activity. The subject will be instructed to grip maximally upon hearing an audible tone. The subject should then relax his/her grip as quickly as possible after hearing a second tone. The relaxation time is defined as the elapsed time in Second from the second tone to the point at which the flexor muscle magnitude returns to the baseline level + three standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Background] Haggard P, Wing A. Coordinated responses following mechanical perturbation of the arm during prehension. Exp Brain Res. 1995;102(3):483-94. doi: 10.1007/BF00230652. PMID 7737394
- [Background] Hoffmann G, Schmit BD, Kahn JH, Kamper DG. Effect of sensory feedback from the proximal upper limb on voluntary isometric finger flexion and extension in hemiparetic stroke subjects. J Neurophysiol. 2011 Nov;106(5):2546-56. doi: 10.1152/jn.00522.2010. Epub 2011 Aug 10. PMID 21832028
- [Background] Kamper DG, Harvey RL, Suresh S, Rymer WZ. Relative contributions of neural mechanisms versus muscle mechanics in promoting finger extension deficits following stroke. Muscle Nerve. 2003 Sep;28(3):309-18. doi: 10.1002/mus.10443. PMID 12929190
- [Background] Kamper DG, Rymer WZ. Quantitative features of the stretch response of extrinsic finger muscles in hemiparetic stroke. Muscle Nerve. 2000 Jun;23(6):954-61. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-0. PMID 10842274
- [Background] Mayer NH, Esquenazi A, Childers MK. Common patterns of clinical motor dysfunction. Muscle Nerve Suppl. 1997;6:S21-35. PMID 9826981
- [Background] Shumway-Cook A, Woollacott MH (2001) Motor Control: Theory and Practical Applications, 2nd ed. vol. Chapter 6. Philadelphia: Lippincott Williams & Wilkins.
- [Background] Ren Y, Kang SH, Park HS, Wu YN, Zhang LQ. Developing a multi-joint upper limb exoskeleton robot for diagnosis, therapy, and outcome evaluation in neurorehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2013 May;21(3):490-9. doi: 10.1109/TNSRE.2012.2225073. Epub 2012 Oct 19. PMID 23096119
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Zhang LQ, Son J, Park HS, Kang SH, Lee Y, Ren Y. Changes of Shoulder, Elbow, and Wrist Stiffness Matrix Post Stroke. IEEE Trans Neural Syst Rehabil Eng. 2017 Jul;25(7):844-851. doi: 10.1109/TNSRE.2017.2707238. Epub 2017 May 23. PMID 28541901
- [Background] Zhang LQ, Xu D, Kang SH, Roth EJ, Ren Y. Multi-Joint Somatosensory Assessment in Patients Post Stroke. BMES Ann Meeting, Phoenix. 2017.